CLINICAL TRIAL: NCT03129061
Title: A Pilot Study to Evaluate Immunological Response to PD-1 Inhibition in Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Study to Evaluate Immunological Response to PD-1 Inhibition in Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CellSight Technologies, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 40425; ENT0061 (Other: Stanford University)
Record Dates: First submitted 2017-04-18; First posted 2017-04-26 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 Patients with M/R SCCHN (Experimental): Patients with unresectable and metastatic SCCHN cancer who will receive anti-PD-1 treatment under SOC. SOC treatments currently include nivolumab and pembrolizumab ("anti-PD-1 treatment"). The protocol may be amended to include other agents should they become SOC. Patients will receive a baseline [18F]F-AraG PET/CT scan and another [18F]F-AraG PET/CT scan 6 to 12 weeks after anti-PD-1 dose.
  Interventions: Drug: [18F]F-AraG PET Scan, baseline + post anti-PD-1 therapy.
- Cohort 2 Patients with de novo SCCHN (Experimental): Patients with de novo SCCHN prior to initiation of anti-cancer treatment (e.g., radiation, chemoradiation, or surgery). Patients will receive ONE DOSE of the anti-PD-1 treatment, after the baseline [18F]F-AraG PET/CT scan, baseline blood and tumor tissue collection. Patients will receive a second [18F]F-AraG PET/CT scan 2 - 3 weeks after the one dose of anti-PD-1 treatment.
  Interventions: Drug: [18F]F-AraG PET Scan, baseline + post anti-PD-1 therapy.

INTERVENTIONS:
Drug: [18F]F-AraG PET Scan, baseline + post anti-PD-1 therapy. — * Baseline: Blood sampling, tumor biopsy, [18F]F-AraG PET/CT scan within two weeks prior to standard of care anti-PD-1 therapeutic dose.
  * Anti PD-1 per standard of care
  * Blood sampling and tumor biopsy within 2-3 weeks after first anti-PD-1 SOC dose.
  * [18F]F-AraG PET/CT scan 6 - 12 weeks post first anti-PD-1 dose.
  Arms: Cohort 1 Patients with M/R SCCHN
Drug: [18F]F-AraG PET Scan, baseline + post anti-PD-1 therapy. — * Baseline: Blood sampling, tumor biopsy, [18F]F-AraG PET/CT scan within two weeks prior to treatment.
  * Anti PD-1, single dose
  * Blood sampling, tumor biopsy and [18F}F-AraG PET/CT scan within 2-3 weeks after single dose of anti-PD-1 treatment. For patients having surgical resection, biopsy will be immediately prior to resection or from sample of resection.
  Arms: Cohort 2 Patients with de novo SCCHN

SUMMARY:
This is a single-center cross-sectional imaging and correlative biomarker study in patients with Squamous Cell Carcinoma of the Head and Neck (SCCHN). Cohort 1 will be patients with unresectable or metastatic SCCHN cancer receiving standard of care (SOC) anti-PD-1 treatment and Cohort 2 will be neoadjuvant study participants who will receive one dose of anti-PD-1 treatment prior to tumor resection or radiation. Blood sampling and tissue biopsies will be collected from both cohorts and both cohorts will undergo two whole body PET(Positron Emission Tomography)/CT(Computed Tomography) imaging with [18F]F-AraG. First scan prior to initiating anti-PD-1 treatment and second scan post initiation of anti-PD-1 treatment in Cohort 1 and prior to tumor resection or radiation in Cohort 2

DETAILED DESCRIPTION:
This is a single-center cross-sectional imaging and correlative biomarker study in patients with Squamous Cell Carcinoma of the Head and Neck (SCCHN). Cohort 1 will be patients with unresectable or metastatic SCCHN cancer receiving standard of care (SOC) anti-PD-1 treatment and cohort 2 will be neoadjuvant study participants who will receive one dose of anti-PD-1 treatment prior to tumor resection or radiation. Blood sampling and tissue biopsies will be collected from both cohorts and both cohorts will undergo two whole body PET(Positron Emission Tomography)/CT(Computed Tomography) imaging with [18F]F-AraG. First scan prior to initiating anti-PD-1 treatment and second scan 6-12 weeks post initiation of anti-PD-1 treatment in Cohort1 and within 2-3 weeks of administration of one dose of anti-PD-1 in Cohort 2.

This study will help us assess if [18F]F-AraG can be used for noninvasive imaging and assessment of T cell activation and expansion in the tumor microenvironment. Specifically, we will be assessing if there is a correlation between an increase in the imaging signal and an increase in T cell activation (measured directly from the T cells obtained from biopsy specimens).

Patients and care providers will not be blinded to any part of this study. Patients will be evaluated one day and one week via telephone visit after each radiopharmaceutical injection for safety follow-up. All adverse events will be recorded. Due to the noninvasive and non-therapeutic nature of the study, potential risks of the study are anticipated to be low.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic SCCHN.
* Localized SCCHN.
* >18 years old.
* Willing and able to sign consent form.
* Have standard of care biopsy or resection planned or tumors amenable to serial biopsies.
* For patients with reproductive potential must undergo counseling to understand unknown risks to resultant progeny.

Exclusion Criteria:

* Diagnosis of immunodeficiency or active autoimmune condition.
* Active tuberculosis
* Prior exposure to PD-1 or PD-LI treatment
* Prior systemic chemotherapy within 2 weeks of planed anti-PD1 treatment.
* Received a live vaccine within 30 days of planned PD-1 start date.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Non-invasive assessment of T cell activation at tumor site from anti-PD1 therapy as measured by signal changes with VisAcT imaging biomarker | Baseline and 6 to 12 weeks after initial anti-PD-1 dose in Cohort 1 and Baseline and 2 to 3 weeks after anti-PD-1 dose in Cohort 2.
  Assess whether [18F]F-AraG accumulation at the site of inflammation can be used for noninvasive imaging and assessment of T cell activation and expansion in the tumor microenvironment. Specifically, we will be assessing if there is a correlation between an increase in the imaging signal and an increase in T cell activation (measured directly from the T cells obtained from biopsy specimens).

SECONDARY OUTCOMES:
Success rate for collection of paired blood and tissue samples pre and post immunotherapy treatment in each Cohort. | 2 to 3 weeks post initial anti-PD-1 dose.
  Explore the feasibility of deep sequencing the tumor cells and also the paired T cell receptor alpha and beta chains of the expanding T cells from the same patient before and after the administration of a Moab directed against PD-1.

CONTACTS AND LOCATIONS:
Overall Officials: A. Dimitrios Colevas, MD, Study Director — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No